CLINICAL TRIAL: NCT07283198
Title: A Phase II Clinical Study to Evaluate the Safety, Efficacy, Pharmacokinetics/Pharmacodynamics of JSKN033 in Patients With Advanced Non-Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JSKN033-201
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Non Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Part 1 (Dose Selection) and Part 2 (Cohort Expansion) (Experimental): JSKN033 is administered at the predefined dose, once per treatment cycle.
  Interventions: Drug: JSKN033 Injection

INTERVENTIONS:
Drug: JSKN033 Injection — JSKN033 is a fixed-dose combination consisting of JSKN003 (a HER2-targeted ADC) and envafolimab (a PD-L1 inhibitor)

SUMMARY:
This is an open-label, multicenter, Phase II clinical study designed to evaluate the safety and efficacy of JSKN033 in the treatment of patients with advanced NSCLC. The study is divided into two phases: Part 1 (Dose Selection) and Part 2 (Cohort Expansion). Enrolled subjects are patients with locally advanced (Stage IIIB/IIIC) or metastatic (Stage IV) NSCLC who are not eligible for curative treatment. Part 1 (Dose Selection): It consists of two dose groups, with a maximum of 20 subjects enrolled in each group. Part 2 (Cohort Expansion): It consists of two cohorts, with a maximum of 60 subjects enrolled in each cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects can understand the informed consent form,voluntarily participate in the study, and sign the informed consent form.
2. Subjects are≥18 years old on the day of signing the informed consent form, regardless of gender.
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
4. Expected survival time ≥3 months.
5. Histologically or cytologically confirmed locally advanced or metastatic NSCLC (per AJCC 8th Edition Lung Cancer TNM Staging) that is not eligible for curative surgery and/or curative radiotherapy.
6. NSCLC confirmed to be no other known driver gene alterations for which first- line targeted therapy has been approved.
7. For Part 1(Dose Selection): Enrolled subjects are those with advanced unresectable or metastatic NSCLC who have failed or are intolerant to standard previous treatments, and have HER2 mutation or HER2 expression in tumor tissue.
8. For Part 2 (Cohort Expansion): Enrolled subjects are those with locally advanced or metastatic NSCLC who have not received prior systemic anti-tumor treatment for their advanced disease.
9. Per RECIST 1.1 criteria,subjects have at least one extracranial measurable lesion at baseline.
10. Subjects must provide tumor tissue samples.
11. Sufficient organ function.
12. Female subjects of childbearing potential or male subjects whose partners are of childbearing potential agree to use highly effective contraceptive measures from the time of signing the informed consent form until 24 weeks after the last dose.

Exclusion Criteria:

1. Presence of any small cell carcinoma component in the histological pathology.
2. History of other malignant tumors within 5 years prior to the first dose administration.
3. History of brainstem, meningeal, or spinal cord metastases/compression, or carcinomatous meningitis; presence of active brain metastases.
4. Imaging during the screening phase shows tumor invasion, compression, or location in surrounding vital organs.
5. Sufficient washout period from previous treatments prior to the first dose.
6. Presence of the following lung diseases or medical history leading to severe respiratory impairment.
7. Presence of risk factors related to interstitial lung disease (ILD) or non-infectious pneumonia.
8. Presence of cardiovascular and cerebrovascular diseases or risk factors.
9. Presence of uncontrolled infections.
10. Toxicity from previous anti-tumor treatment has not recovered to grade≤1 (per CTCAE v5.0).
11. Previous history of allogeneic bone marrow or organ transplantation.
12. Known allergy to any component of the study drug.
13. Pregnant and/or lactating women, or women planning to become pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Number and Severity of Treatment-emergent Adverse Events (TEAEs) | Baseline up to 30 days after the last dose of study drug, up to 1 year
  The incidence and severity of TEAEs and TRAEs (Treatment-related Adverse Events, graded according to NCI CTCAE 5.0), Serious AEs (SAEs), laboratory tests, etc.
Objective response rate (ORR) | Up to 1 year after the last participant receives the last dose
  ORR was defined as the proportion of subjects achieving Complete Response (CR) or Partial Response (PR)

SECONDARY OUTCOMES:
Duration of response (DoR) | Up to 1 year after the last participant receives the last dose
  Duration of response for responders (CR or PR) is defined as the time interval between the date of earliest qualifying response and the date of PD or death for any cause, whichever occurs earlier
Disease control rate (DCR) | Up to 1 year after the last participant receives the last dose
  DCR was defined as the proportion of subjects whose best overall response is CR, PR, or Stable Disease (SD)
Clinical benefit rate (CBR) | Up to 1 year after the last participant receives the last dose
  Clinical benefit rate (CR+PR+[stable disease (SD) ≥ 6 months]) is defined as those participants with best response as CR or PR or else SD with a duration of at least 6 months. SD for 6 months duration was defined as the time from the first dose to the first documentation of PD or to the last adequate response assessment prior to data cut-off date, whichever is earlier.
Progression-free Survival (PFS) | Up to 1 year after the last participant receives the last dose
  PFS is defined as the time from the date of first study dose to disease progression or death whichever occurs first. Subjects without event (no disease progression or alive at last visit) will be censored at the date of "last tumor assessment".
Overall survival (OS) | Up to 1 year after the last participant receives the last dose
  OS was defined as the time from the date of first dose until the date of death from any cause
PK parameter: Cmax | Post last dose up to Day 90
  Maximum (Peak) Observed blood Concentration (Cmax)
PK parameter: Tmax | Post last dose up to Day 90
  Time of Maximum blood Concentration (Tmax)
PK parameter: AUC | Post last dose up to Day 90
  The blood PK parameters of JSKN033 and its analytes for area under the concentration-versus-time curve from time 0 to the last quantifiable concentration as calculated by the linear-up log-down trapezoidal method (AUClast) and AUC from time 0 to infinity (AUCinf) elimination rate constant associated with the terminal phase were estimated using standard non-compartmental methods.
PK parameter: Terminal Elimination Half-life (t1/2) | Post last dose up to Day 90
PK parameter: Volume of distribution (V) | Post last dose up to Day 90
PK parameter: trough concentration (Ctrough) | Post last dose up to Day 90
PK parameter: Clearance (CL) | Post last dose up to Day 90
PK parameter: Accumulation index (Rac) | Post last dose up to Day 90
PK parameter: Mean residence time (MRT) | Post last dose up to Day 90
Incidence of anti-drug antibodies (ADAs), antibody titers, and incidence of neutralizing antibodies | Post last dose up to Day 90

OTHER OUTCOMES:
Correlation between biomarkers (HER2 mutation status, HER2/PD-L1 expression levels) in tumor tissue samples and efficacy. | Up to 1 year after the last participant receives the last dose

IPD SHARING:
Plan to Share IPD: Undecided